CLINICAL TRIAL: NCT01229436
Title: Prospective Open-Label Investigation Of The Non-surgical Treatment With Collagenase Clostridium Histolyticum (Xiapex)
Brief Title: Treatment Of Dupuytren's Contracture With Collagenase Clostridium Histolyticum Injection (Xiapex)
Acronym: POINT X
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1531002
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-01

CONDITIONS: Dupuytren's Contracture
Keywords: Dupuytren's; treatment; injection; recovery; health care resources
MeSH Terms: conditions — Dupuytren Contracture | interventions — xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xiapex Injection (Experimental)
  Interventions: Drug: Xiapex

INTERVENTIONS:
Drug: Xiapex — Xiapex 0.58 mg in diluent, 0.25 ml for MP joints and 0.20 ml for PIP joints, injection to cord over joint using either 26 or 27 gauge needle, maximum 3 injections with 30 days interval between injections to any single site, maximum 5 injections in this protocol

SUMMARY:
This study will evaluate the impact of Xiapex treatment on the range of motion (ROM) of the affected fingers and the patient and physician reported treatment satisfaction and disease severity and their relation to ROM. Recovery to normal activities, recovery time (How long overall, time to use hand, time to return to work or daily activities, amount of work or daily activity time missed or reduced and affects on productivity and daily activities) will be assessed via patient diary. Use of concomitant analgesic medications will be recorded and total healthcare resource utilization (HCRU).

ELIGIBILITY:
Inclusion Criteria:

* Presenting with a Dupuytren's contracture of at least 20 degrees caused by a palpable cord in at least one finger other than the thumb.
* Positive "table top test" defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top.

Exclusion Criteria:

* Received a treatment on the selected joint, within 90 days of enrollment in the study, for Dupuytren's contracture including needle aponeurotomy or any surgical procedure
* On anticoagulant medication or has received anticoagulant medication (except aspirin less than 150 mg daily) within 7 days before the first injection
* Has a chronic muscular, neurological, or neuromuscular disorder that affects the hands

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Denmark (2):
  - Pfizer Investigational Site, Copenhagen
  - Pfizer Investigational Site, Silkeborg
- France (3):
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
- Germany (6):
  - Pfizer Investigational Site, Bad Neustadt an der Saale
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Tübingen
- Pfizer Investigational Site, Miskolc, Hungary
- Italy (3):
  - Pfizer Investigational Site, Sesto San Giovanni, Milano
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Savona
- Spain (5):
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona/ Spain
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Málaga, Málaga
  - Pfizer Investigational Site, Barcelona
- Sweden (3):
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- United Kingdom (4):
  - Pfizer Investigational Site, Derby
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Norwich
  - Pfizer Investigational Site, Southampton

REFERENCES:
- [Derived] Warwick D, Arner M, Pajardi G, Reichert B, Szabo Z, Masmejean EH, Fores J, Chapman DS, Gerber RA, Huard F, Seghouani A, Szczypa PP; POINT X Investigators. Collagenase clostridium histolyticum in patients with Dupuytren's contracture: results from POINT X, an open-label study of clinical and patient-reported outcomes. J Hand Surg Eur Vol. 2015 Feb;40(2):124-32. doi: 10.1177/1753193413519926. Epub 2014 Jan 26. PMID 24470559
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1531002&StudyName=Treatment%20Of%20Dupuytren%27s%20Contracture%20With%20Collagenase%20Clostridium%20Histolyticum%20Injection%20%28Xiapex%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Xiapex: A single injection of Xiapex (collagenase clostridium histolyticum) 0.58 milligram (mg) directly into the cord over metacarpophalangeal (MP) joint or proximal interphalangeal (PIP) joint of a finger on injection day followed by a finger extension procedure and 30-day follow-up period in each cycle up to 5 cycles. A maximum of 3 injections were allowed into a single cord. Participants were followed-up at Day 90 and 180 after the last treatment cycle.
Period: Overall Study
Arm/Group | Xiapex
Started | 254
Completed | 249
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 223

OUTCOME MEASURES:

1. Primary Outcome: Total Passive Extension Deficit (TPED) at Baseline for First Injection
Description: TPED was defined as the sum of passive extension deficits (PED) in the MP, PIP and distal interphalangeal (DIP) joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. Baseline value for first injection was the TPED value taken closest and prior to the administration of first injection. Baseline value after first injection was also considered as baseline for follow-up on Day 90, 180 after last injection (follow-up baseline). 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Baseline for first injection
Population: Full analysis set(FAS):participants who received at least (>=)1 injection of Xiapex,had >=1 post-injection efficacy assessment(goniometric/participant-reported). 'N'(number of participants analyzed) includes total number of participants in FAS, however actual 'N' for this outcome is unknown as these data were not calculated as per planned analysis.
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 259
degrees | 55.0 [2 to 180]

2. Secondary Outcome: Passive Extension Deficit (PED) for Metacarpophalangeal (MP) and Proximal Interphalangeal (PIP) Joints
Description: PED was measured in MP and PIP joints using finger goniometry. Passive extension=angle of the joint (MP or PIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. For each injection, baseline value was the PED value taken closest and prior to administration of that particular injection. For follow-up on Day 90 and 180 after last injection, baseline value (follow-up baseline) was the PED value taken closest and prior to administration of first injection in that joint. PED was reported at Day 1, 7 and 30 after each injection for joints that received 1 through 3 injections and at Day 90 and 180 after the last injection, where last injection was a maximum up to third injection for a joint. 'Number of joints analyzed' signifies total number of MP and PIP joints analyzed for this outcome measure and 'n' signifies number of joints evaluable for this measure at given time points for the mentioned joint.
Time Frame: Baseline for first, second, third injection; Day 1, 7, 30 after first, second, third injection; Follow-up: Day 90, 180 after last injection
Population: FAS: participants who received >=1 injection of Xiapex, had >=1 post-injection efficacy assessment, whether goniometric or participant-reported. 'N' (number of participants analyzed) includes total number of participants in FAS, however actual 'N' for this outcome is unknown as these data were not calculated as per planned analysis.
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Joints) | 309
degrees
  Baseline for first injection: MP Joint (n=211) | 40.0 [0 to 90]
  Day 1 after first injection: MP Joint (n=207) | 8.0 [0 to 80]
  Day 7 after first injection: MP Joint (n=209) | 0.0 [0 to 82]
  Day 30 after first injection: MP Joint (n=209) | 0.0 [0 to 70]
  Baseline for second injection: MP Joint (n=33) | 25.0 [0 to 74]
  Day 1 after second injection: MP Joint (n=33) | 5.0 [0 to 45]
  Day 7 after second injection: MP Joint (n=33) | 5.0 [0 to 50]
  Day 30 after second injection: MP Joint (n=32) | 8.5 [0 to 30]
  Baseline for third injection: MP Joint (n=9) | 20.0 [0 to 50]
  Day 1 after third injection: MP Joint (n=9) | 0.0 [0 to 50]
  Day 7 after third injection: MP Joint (n=9) | 10.0 [0 to 40]
  Day 30 after third injection: MP Joint (n=9) | 20.0 [0 to 40]
  Baseline for follow-up: MP Joint (n=201) | 40.0 [0 to 90]
  Follow-up Day 90: MP Joint (n=201) | 0.0 [0 to 70]
  Follow-up Day 180: MP Joint (n=207) | 0.0 [0 to 85]
  Baseline for first injection: PIP Joint (n=98) | 45.0 [15 to 94]
  Day 1 after first injection: PIP Joint (n=98) | 20.0 [0 to 80]
  Day 7 after first injection: PIP Joint (n=97) | 14.0 [0 to 90]
  Day 30 after first injection: PIP Joint (n=98) | 18.5 [0 to 90]
  Baseline for second injection: PIP Joint (n=18) | 40.0 [5 to 90]
  Day 1 after second injection: PIP Joint (n=15) | 30.0 [0 to 90]
  Day 7 after second injection: PIP Joint (n=18) | 30.0 [0 to 90]
  Day 30 after second injection: PIP Joint (n=18) | 27.0 [0 to 95]
  Baseline for third injection: PIP Joint (n=6) | 37.5 [20 to 80]
  Day 1 after third injection: PIP Joint (n=6) | 12.5 [0 to 70]
  Day 7 after third injection: PIP Joint (n=6) | 17.5 [0 to 80]
  Day 30 after third injection: PIP Joint (n=6) | 20.0 [5 to 80]
  Baseline for follow-up: PIP Joint (n=93) | 45.0 [15 to 94]
  Follow-up Day 90: PIP Joint (n=93) | 20.0 [0 to 80]
  Follow-up Day 180: PIP Joint (n=93) | 25.0 [0 to 80]

3. Secondary Outcome: Change From Baseline in Total Passive Extension Deficit (TPED) at Day 1, 7 and 30 After First, Second, Third and Fourth Injection, Day 90 and 180 After Last Injection
Description: TPED was defined as sum of PED in MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. For each injection, baseline value was TPED value taken closest and prior to administration of that particular injection. Baseline value after first injection was also considered as baseline for follow-up on Day 90, 180 after last injection (follow-up baseline). Change in TPED was reported at Day 1, 7 and 30 after each injection for fingers that received 1 through 4 injections and at Day 90, 180 after last injection, where last injection was a maximum up to fourth injection for a finger. Results are not reported for fifth injection as no finger received 5 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Baseline for first, second, third, fourth injection; Day 1, 7, 30 after first, second, third, fourth injection; Follow-up Day 90, 180 after last injection
Population: FAS population. 'N' (number of participants analyzed) includes total number of participants in FAS,however actual 'N' for this outcome is unknown as these data were not calculated as per planned analysis. Here, 'n' signifies number of fingers/joints evaluable for this outcome measure at given time points.
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 257
degrees
  Change at Day 1 after first injection (n=256) | -31.0 [-145 to 35]
  Change at Day 7 after first injection (n=256) | -40.0 [-160 to 15]
  Change at Day 30 after first injection (n=257) | -40.0 [-155 to 7]
  Change at Day 1 after second injection (n=64) | -20.0 [-85 to 33]
  Change at Day 7 after second injection (n=65) | -20.0 [-85 to 31]
  Change at Day 30 after second injection (n=64) | -20.0 [-89 to 31]
  Change at Day 1 after third injection (n=19) | -15.0 [-45 to 3]
  Change at Day 7 after third injection (n=21) | -10.0 [-45 to 20]
  Change at Day 30 after third injection (n=21) | -10.0 [-20 to 20]
  Change at Day 1 after fourth injection (n=1) | -20.0 [-20 to -20]
  Change at Day 7 after fourth injection (n=1) | -20.0 [-20 to -20]
  Change at Day 30 after fourth injection (n=1) | -10.0 [-10 to -10]
  Change at Follow-up Day 90 (n=244) | -40.0 [-155 to 25]
  Change at Follow-up Day 180 (n=250) | -35.0 [-165 to 50]

4. Secondary Outcome: Change From Baseline in Passive Extension Deficit (PED) for Metacarpophalangeal (MP) and Proximal Interphalangeal (PIP) Joints at Day 1, 7 and 30 After First, Second and Third Injection, Day 90 and 180 After Last Injection
Description: PED was measured in MP and PIP joints using finger goniometry. Passive extension=angle of the joint (MP or PIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. For each injection, baseline value was the PED value taken closest and prior to administration of that particular injection. For follow-up on Day 90 and 180 after last injection, baseline value (follow-up baseline) was the PED value taken closest and prior to administration of first injection in that joint. Change in PED was reported at Day 1, 7 and 30 after each injection for joints that received 1 through 3 injections and at Day 90 and 180 after the last injection, where last injection was a maximum up to third injection for a joint. 'Number of joints analyzed' signifies total number of MP and PIP joints analyzed for this outcome measure and 'n' signifies number of joints evaluable for this measure at given time points for the mentioned joint.
Time Frame: Baseline for first, second, third injection; Day 1, 7, 30 after first, second, third injection; Follow-up Day 90, 180 after last injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Joints) | 307
degrees
  Change at Day 1 after first injection: MP(n=207) | -30.0 [-90 to 25]
  Change at Day 7 after first injection: MP(n=209) | -30.0 [-80 to 12]
  Change at Day 30 after first injection: MP(n=209) | -35.0 [-80 to 10]
  Change at Day 1 after second injection: MP(n=33) | -20.0 [-60 to 10]
  Change at Day 7 after second injection: MP(n=33) | -20.0 [-58 to 20]
  Change at Day 30 after second injection: MP(n=32) | -20.0 [-68 to 10]
  Change at Day 1 after third injection: MP(n=9) | -10.0 [-30 to 0]
  Change at Day 7 after third injection: MP(n=9) | -10.0 [-30 to 10]
  Change at Day 30 after third injection: MP(n=9) | -10.0 [-10 to 10]
  Change at Follow-up Day 90: MP(n=201) | -35.0 [-88 to 10]
  Change at Follow-up Day 180: MP(n=207) | -35.0 [-82 to 20]
  Change at Day 1 after first injection: PIP(n=98) | -25.0 [-90 to 33]
  Change at Day 7 after first injection: PIP(n=97) | -30.0 [-90 to 31]
  Change at Day 30 after first injection: PIP(n=98) | -30.0 [-94 to 31]
  Change at Day 1 after second injection: PIP(n=15) | -10.0 [-42 to 6]
  Change at Day 7 after second injection: PIP(n=18) | -12.5 [-45 to 6]
  Change at Day 30 after second injection: PIP(n=18) | -14.5 [-40 to 10]
  Change at Day 1 after third injection: PIP(n=6) | -20.0 [-30 to 0]
  Change at Day 7 after third injection: PIP(n=6) | -16.5 [-35 to 0]
  Change at Day 30 after third injection: PIP(n=6) | -15.0 [-20 to 0]
  Change at Follow-up Day 90: PIP(n=93) | -20.0 [-90 to 25]
  Change at Follow-up Day 180: PIP(n=93) | -20.0 [-94 to 25]

5. Secondary Outcome: Range of Motion (ROM) for Metacarpophalangeal (MP) and Proximal Interphalangeal (PIP) Joints
Description: Finger goniometry was used to measure the angles of extension and flexion of MP and PIP joints. ROM was measured as the difference between the angle of flexion and the angle of extension of the joint. For each injection, baseline value was the ROM value taken closest and prior to administration of that particular injection. For follow-up on Day 90 and 180 after last injection, baseline value (follow-up baseline) was the ROM value taken closest and prior to administration of first injection in that joint. ROM was reported at Day 1, 7 and 30 after each injection for joints that received 1 through 3 injections and at Day 90 and 180 after the last injection, where last injection was a maximum up to third injection for a joint. 'Number of joints analyzed' signifies total number of MP and PIP joints analyzed for this outcome measure and 'n' signifies number of joints evaluable for this measure at given time points for the mentioned joint.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Joints) | 307
degrees
  Baseline for first injection: MP Joint (n=208) | 45.0 [0 to 90]
  Day 1 after first injection: MP Joint (n=207) | 65.0 [10 to 90]
  Day 7 after first injection: MP Joint (n=209) | 80.0 [-42 to 105]
  Day 30 after first injection: MP Joint (n=209) | 86.0 [20 to 105]
  Baseline for second injection: MP Joint (n=33) | 60.0 [10 to 90]
  Day 1 after second injection: MP Joint (n=33) | 76.0 [20 to 90]
  Day 7 after second injection: MP Joint (n=32) | 80.0 [6 to 95]
  Day 30 after second injection: MP Joint (n=32) | 80.0 [28 to 95]
  Baseline for third injection: MP Joint (n=9) | 70.0 [40 to 90]
  Day 1 after third injection: MP Joint (n=9) | 90.0 [40 to 90]
  Day 7 after third injection: MP Joint (n=9) | 80.0 [45 to 90]
  Day 30 after third injection: MP Joint (n=9) | 70.0 [50 to 90]
  Baseline for follow-up: MP Joint (n=198) | 45.0 [0 to 90]
  Follow-up Day 90: MP Joint (n=201) | 90.0 [20 to 110]
  Follow-up Day 180: MP Joint (n=207) | 90.0 [10 to 110]
  Baseline for first injection: PIP Joint (n=98) | 50.0 [0 to 85]
  Day 1 after first injection: PIP Joint (n=98) | 63.0 [10 to 100]
  Day 7 after first injection: PIP Joint (n=97) | 75.0 [10 to 110]
  Day 30 after first injection: PIP Joint (n=98) | 75.5 [10 to 105]
  Baseline for second injection: PIP Joint (n=18) | 50.0 [10 to 85]
  Day 1 after second injection: PIP Joint (n=15) | 50.0 [10 to 90]
  Day 7 after second injection: PIP Joint (n=18) | 67.0 [20 to 90]
  Day 30 after second injection: PIP Joint (n=18) | 65.0 [10 to 90]
  Baseline for third injection: PIP Joint (n=6) | 57.5 [10 to 70]
  Day 1 after third injection: PIP Joint (n=6) | 80.0 [20 to 90]
  Day 7 after third injection: PIP Joint (n=6) | 80.0 [10 to 90]
  Day 30 after third injection: PIP Joint (n=6) | 72.5 [10 to 85]
  Baseline for follow-up: PIP Joint (n=93) | 50.0 [0 to 85]
  Follow-up Day 90: PIP Joint (n=93) | 72.0 [10 to 105]
  Follow-up Day 180: PIP Joint (n=93) | 70.0 [10 to 105]

6. Secondary Outcome: Participant Global Assessment of Treatment Satisfaction and Disease Severity
Description: Participant global assessment questionnaire assessed severity of the contracture at baseline, post-injection and treatment satisfaction (TS), improvement from baseline in the treated contracture at post-injection only. Participants rated disease severity as normal (no contracture), mild, moderate or severe. Overall satisfaction was rated as very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied or very dissatisfied. Participants rated their improvement in disease severity relative to baseline on a 11-point scale ranging from 0 percent (%) = no improvement to 100% = total recovery, with 10 % increment between each point. Results are reported for number of participants in each category for disease severity, TS and improvement.
Time Frame: Baseline for cycle 1, 2, 3, 4, 5; Cycle 1 Day 30 (C1D30), C2D30, C3D30, C4D30, C5D30; Follow-up (FU) Day 90, 180 after last injection
Population: FAS: participants who received >= 1 injection of Xiapex, had >=1 post-injection efficacy assessment, whether goniometric or participant-reported. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: participants
Arm/Group | Xiapex
Number analyzed (Participants) | 254
participants
  Baseline for cycle 1, severity: normal (n=254) | 2
  Baseline for cycle 1, severity: mild (n=254) | 40
  Baseline for cycle 1, severity: moderate (n=254) | 128
  Baseline for cycle 1, severity: severe (n=254) | 84
  C1D30, severity: normal (n=253) | 63
  C1D30, severity: mild (n=253) | 114
  C1D30, severity: moderate (n=253) | 55
  C1D30, severity: severe (n=253) | 21
  C1D30, TS: very satisfied (n=253) | 153
  C1D30, TS: satisfied (n=253) | 73
  C1D30, TS: neither satisfied/dissatisfied (n=253) | 16
  C1D30, TS: dissatisfied (n=253) | 6
  C1D30, TS: very dissatisfied (n=253) | 5
  C1D30, improvement: 0% (n=252) | 10
  C1D30, improvement: 10% (n=252) | 11
  C1D30, improvement: 20% (n=252) | 6
  C1D30, improvement: 30% (n=252) | 8
  C1D30, improvement: 40% (n=252) | 6
  C1D30, improvement: 50% (n=252) | 20
  C1D30, improvement: 60% (n=252) | 15
  C1D30, improvement: 70% (n=252) | 19
  C1D30, improvement: 80% (n=252) | 52
  C1D30, improvement: 90% (n=252) | 58
  C1D30, improvement: 100% (n=252) | 47
  Baseline for cycle 2, severity: mild (n=112) | 22
  Baseline for cycle 2, severity: moderate (n=112) | 62
  Baseline for cycle 2, severity: severe (n=112) | 28
  C2D30, severity: normal (n=109) | 27
  C2D30, severity: mild (n=109) | 47
  C2D30, severity: moderate (n=109) | 24
  C2D30, severity: severe (n=109) | 11
  C2D30, TS: very satisfied (n=109) | 64
  C2D30, TS: satisfied (n=109) | 37
  C2D30, TS: neither satisfied/dissatisfied (n=109) | 6
  C2D30, TS: dissatisfied (n=109) | 1
  C2D30, TS: very dissatisfied (n=109) | 1
  C2D30, improvement: 0% (n=109) | 4
  C2D30, improvement: 10% (n=109) | 1
  C2D30, improvement: 20% (n=109) | 2
  C2D30, improvement: 30% (n=109) | 7
  C2D30, improvement: 40% (n=109) | 4
  C2D30, improvement: 50% (n=109) | 10
  C2D30, improvement: 60% (n=109) | 9
  C2D30, improvement: 70% (n=109) | 8
  C2D30, improvement: 80% (n=109) | 13
  C2D30, improvement: 90% (n=109) | 33
  C2D30, improvement: 100% (n=109) | 18
  Baseline for cycle 3, severity: normal (n=54) | 1
  Baseline for cycle 3, severity: mild (n=54) | 14
  Baseline for cycle 3, severity: moderate (n=54) | 25
  Baseline for cycle 3, severity: severe (n=54) | 14
  C3D30, severity: normal (n=54) | 8
  C3D30, severity: mild (n=54) | 26
  C3D30, severity: moderate (n=54) | 16
  C3D30, severity: severe (n=54) | 4
  C3D30, TS: very satisfied (n=54) | 29
  C3D30, TS: satisfied (n=54) | 18
  C3D30, TS: neither satisfied/dissatisfied (n=54) | 4
  C3D30, TS: dissatisfied (n=54) | 3
  C3D30, improvement: 0% (n=54) | 2
  C3D30, improvement: 10% (n=54) | 1
  C3D30, improvement: 20% (n=54) | 1
  C3D30, improvement: 30% (n=54) | 3
  C3D30, improvement: 40% (n=54) | 2
  C3D30, improvement: 60% (n=54) | 7
  C3D30, improvement: 70% (n=54) | 11
  C3D30, improvement: 80% (n=54) | 8
  C3D30, improvement: 90% (n=54) | 16
  C3D30, improvement: 100% (n=54) | 3
  Baseline for cycle 4, severity: mild (n=24) | 11
  Baseline for cycle 4, severity: moderate (n=24) | 9
  Baseline for cycle 4, severity: severe (n=24) | 4
  C4D30, severity: normal (n=24) | 2
  C4D30, severity: mild (n=24) | 13
  C4D30, severity: moderate (n=24) | 8
  C4D30, severity: severe (n=24) | 1
  C4D30, TS: very satisfied (n=24) | 13
  C4D30, TS: satisfied (n=24) | 9
  C4D30, TS: dissatisfied (n=24) | 2
  C4D30, improvement: 10% (n=24) | 2
  C4D30, improvement: 20% (n=24) | 1
  C4D30, improvement: 40% (n=24) | 2
  C4D30, improvement: 50% (n=24) | 3
  C4D30, improvement: 60% (n=24) | 3
  C4D30, improvement: 70% (n=24) | 3
  C4D30, improvement: 80% (n=24) | 5
  C4D30, improvement: 90% (n=24) | 2
  C4D30, improvement: 100% (n=24) | 3
  Baseline for cycle 5, severity: mild (n=12) | 7
  Baseline for cycle 5, severity: moderate (n=12) | 4
  Baseline for cycle 5, severity: severe (n=12) | 1
  C5D30, severity: normal (n= 12) | 1
  C5D30, severity: mild (n= 12) | 6
  C5D30, severity: moderate (n= 12) | 4
  C5D30, severity: severe (n= 12) | 1
  C5D30, TS: very satisfied (n= 12) | 8
  C5D30, TS: satisfied (n= 12) | 3
  C5D30, TS: neither satisfied/dissatisfied (n= 12) | 1
  C5D30, improvement: 10% (n= 12) | 1
  C5D30, improvement: 70% (n= 12) | 2
  C5D30, improvement: 80% (n= 12) | 4
  C5D30, improvement: 90% (n= 12) | 5
  FU Day 90, severity: normal (n=246) | 92
  FU Day 90, severity: mild (n=246) | 102
  FU Day 90, severity: moderate (n=246) | 43
  FU Day 90, severity: severe (n=246) | 9
  FU Day 90, TS: very satisfied (n=247) | 163
  FU Day 90, TS: satisfied (n=247) | 57
  FU Day 90,TS:neither satisfied/dissatisfied(n=247) | 10
  FU Day 90, TS: satisfaction: dissatisfied (n=247) | 13
  FU Day 90, TS:very dissatisfied (n=247) | 4
  FU Day 90, improvement: 0% (n=247) | 7
  FU Day 90, improvement: 10% (n=247) | 4
  FU Day 90, improvement: 20% (n=247) | 6
  FU Day 90, improvement: 30% (n=247) | 3
  FU Day 90, improvement: 40% (n=247) | 6
  FU Day 90, improvement: 50% (n=247) | 13
  FU Day 90, improvement: 60% (n=247) | 5
  FU Day 90, improvement: 70% (n=247) | 20
  FU Day 90, improvement: 80% (n=247) | 42
  FU Day 90, improvement: 90% (n=247) | 78
  FU Day 90, improvement: 100% (n=247) | 63
  FU Day 180, severity: normal (n=248) | 78
  FU Day 180, severity: mild (n=248) | 96
  FU Day 180, severity: moderate (n=248) | 54
  FU Day 180, severity: severe (n=248) | 20
  FU Day 180, TS: very satisfied (n=249) | 152
  FU Day 180, TS: satisfied (n=249) | 64
  FU Day180,TS:neither satisfied/dissatisfied(n=249) | 13
  FU Day 180,TS: dissatisfied (n=249) | 15
  FU Day 180,TS: very dissatisfied (n=249) | 5
  FU Day 180, improvement: 0% (n=249) | 17
  FU Day 180, improvement: 10% (n=249) | 5
  FU Day 180, improvement: 20% (n=249) | 2
  FU Day 180, improvement: 30% (n=249) | 4
  FU Day 180, improvement: 40% (n=249) | 4
  FU Day 180, improvement: 50% (n=249) | 15
  FU Day 180, improvement: 60% (n=249) | 6
  FU Day 180, improvement: 70% (n=249) | 21
  FU Day 180, improvement: 80% (n=249) | 43
  FU Day 180, improvement: 90% (n=249) | 74
  FU Day 180, improvement: 100% (n=249) | 58

7. Secondary Outcome: Physician Global Assessment of Treatment Satisfaction and Disease Severity
Description: Physician global assessment questionnaire assessed severity of the contracture at baseline, post-injection and TS, improvement from baseline in the treated contracture at post-injection only. Physician's rated disease severity as normal (no contracture), mild, moderate or severe. Overall satisfaction was rated as very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied or very dissatisfied. Physicians rated participant's improvement in disease severity relative to baseline as very much improved, much improved, minimally improved, no change, minimally worse, much worse or very much worse.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Xiapex
Number analyzed (Participants) | 254
participants
  Baseline for cycle 1, severity: mild (n=254) | 51
  Baseline for cycle 1, severity: moderate (n=254) | 138
  Baseline for cycle 1, severity: severe (n=254) | 65
  C1D30, severity: normal (n=250) | 60
  C1D30, severity: mild (n=250) | 106
  C1D30, severity: moderate (n=250) | 62
  C1D30, severity: severe (n=250) | 22
  C1D30, TS: very satisfied (n=250) | 134
  C1D30, TS: satisfied (n=250) | 90
  C1D30, TS: neither satisfied/dissatisfied (n=250) | 14
  C1D30, TS: dissatisfied (n=250) | 7
  C1D30, TS: very dissatisfied (n=250) | 5
  C1D30, improvement: very much improved (n=250) | 121
  C1D30, improvement: much improved (n=250) | 88
  C1D30, improvement: minimally improved (n=250) | 26
  C1D30, improvement: no change (n=250) | 14
  C1D30, improvement: minimally worse (n=250) | 1
  Baseline for cycle 2, severity: mild (n=110) | 33
  Baseline for cycle 2, severity: moderate (n=110) | 53
  Baseline for cycle 2, severity: severe (n=110) | 24
  C2D30, severity: normal (n=108) | 20
  C2D30, severity: mild (n=108) | 51
  C2D30, severity: moderate (n=108) | 28
  C2D30, severity: severe (n=108) | 9
  C2D30, TS: very satisfied (n=108) | 63
  C2D30, TS: satisfied (n=108) | 36
  C2D30, TS: neither satisfied/dissatisfied (n=108) | 5
  C2D30, TS: dissatisfied (n=108) | 3
  C2D30, TS: very dissatisfied (n=108) | 1
  C2D30,improvement:very much improved (n=108) | 41
  C2D30, improvement:much improved (n=108) | 55
  C2D30, improvement:minimally improved (n=108) | 8
  C2D30, improvement:no change (n=108) | 4
  Baseline for cycle 3, severity: mild (n=53) | 16
  Baseline for cycle 3, severity: moderate (n=53) | 25
  Baseline for cycle 3, severity: severe (n=53) | 12
  C3D30, severity: normal (n=53) | 9
  C3D30, severity: mild (n=53) | 24
  C3D30, severity: moderate (n=53) | 13
  C3D30, severity: severe (n=53) | 7
  C3D30, TS: very satisfied (n=53) | 26
  C3D30, TS: satisfied (n=53) | 22
  C3D30, TS: neither satisfied/dissatisfied (n=53) | 4
  C3D30, TS: dissatisfied (n=53) | 1
  C3D30, improvement: very much improved (n=53) | 22
  C3D30, improvement: much improved (n=53) | 24
  C3D30, improvement: minimally improved (n=53) | 5
  C3D30, improvement: no change (n=53) | 2
  Baseline for cycle 4, severity: mild (n=24) | 10
  Baseline for cycle 4, severity: moderate (n=24) | 9
  Baseline for cycle 4, severity: severe (n=24) | 5
  C4D30, severity: normal (n=24) | 2
  C4D30, severity: mild (n=24) | 11
  C4D30, severity: moderate (n=24) | 8
  C4D30, severity: severe (n=24) | 3
  C4D30, TS: very satisfied (n=24) | 4
  C4D30, TS: satisfied (n=24) | 15
  C4D30, TS: neither satisfied/dissatisfied (n=24) | 1
  C4D30, TS: dissatisfied (n=24) | 1
  C4D30, improvement: very much improved (n=24) | 6
  C4D30, improvement: much improved (n=24) | 14
  C4D30, improvement: minimally improved (n=24) | 3
  C4D30, improvement: no change (n=24) | 1
  Baseline for cycle 5, severity: mild (n=12) | 5
  Baseline for cycle 5, severity: moderate (n=12) | 5
  Baseline for cycle 5, severity: severe (n=12) | 2
  C5D30, severity: mild (n= 12) | 7
  C5D30, severity: moderate (n= 12) | 3
  C5D30, severity: severe (n= 12) | 2
  C5D30, TS: very satisfied (n= 12) | 7
  C5D30, TS: satisfied (n= 12) | 3
  C5D30, TS: neither satisfied/dissatisfied (n= 12) | 2
  C5D30, improvement: very much improved (n=12) | 5
  C5D30, improvement: much improved (n=12) | 5
  C5D30, improvement: minimally improved (n=12) | 1
  C5D30, improvement: no change (n=12) | 1
  FU Day 90, severity: normal (n=247) | 70
  FU Day 90, severity: mild (n=247) | 117
  FU Day 90, severity: moderate (n=247) | 51
  FU Day 90, severity: severe (n=247) | 9
  FU Day 90, TS: very satisfied (n=247) | 145
  FU Day 90, TS: satisfied (n=247) | 75
  FU Day 90,TS:neither satisfied/dissatisfied(n=247) | 15
  FU Day 90, TS: dissatisfied (n=247) | 10
  FU Day 90, TS: very dissatisfied (n=247) | 2
  FU Day 90, improvement: very much improved (n=247) | 123
  FU Day 90, improvement: much improved (n=247) | 95
  FU Day 90, improvement: minimally improved (n=247) | 17
  FU Day 90, improvement: no change (n=247) | 11
  FU Day 90, improvement: much worse (n=247) | 1
  FU Day 180, severity: normal (n=249) | 67
  FU Day 180, severity: mild (n=249) | 114
  FU Day 180, severity: moderate (n=249) | 47
  FU Day 180, severity: severe (n=249) | 21
  FU Day 180, TS: very satisfied (n=249) | 117
  FU Day 180, TS: satisfied (n=249) | 97
  FU Day180,TS:neither satisfied/dissatisfied(n=249) | 15
  FU Day 180, TS: dissatisfied (n=249) | 12
  FU Day 180, TS: very dissatisfied(n=249) | 8
  FU Day 180, improvement:very much improved(n=249) | 94
  FU Day 180, improvement: much improved (n=249) | 114
  FU Day 180, improvement:minimally improved(n=249) | 18
  FU Day 180, improvement:no change (n=249) | 13
  FU Day 180, improvement: minimally worse (n=249) | 5
  FU Day 180, improvement: much worse (n=249) | 4
  FU Day 180, improvement: very much worse (n=249) | 1

8. Secondary Outcome: Number of Participants With Type of Concomitant Pain Medication Used
Description: Number of participants who took different types of analgesic medications, including acetylsalicylic acid, other analgesics (any other analgesic besides those mentioned, as approved by the investigator), aporex, codis, dihydrocodeine, fentanyl, galenic/paracetamol/codeine/, hot coldrex, metamizole, morphine, oxycodone, panadeine CO (combination of paracetamol and codeine phosphate), paracetamol, paramol-118, pregabalin, solpadeine, tramadol, ultracet, to manage pain symptoms were reported. A single participant may be represented in more than 1 category.
Time Frame: Screening up to Day 180 after last injection
Population: Safety set included all participants who received at least 1 injection of Xiapex.
Measure: Number; unit: participants
Arm/Group | Xiapex
Number analyzed (Participants) | 254
participants
  Acetylsalicylic acid | 5
  Other analgesics | 2
  Aporex | 1
  Codis | 1
  Dihydrocodeine | 1
  Fentanyl | 3
  Galenic/Paracetamol/Codeine | 2
  Hot coldrex | 1
  Metamizole | 4
  Morphine | 3
  Oxycodone | 1
  Panadeine CO | 11
  Paracetamol | 96
  Paramol-118 | 1
  Pregabalin | 2
  Solpadeine | 1
  Tramadol | 7
  Ultracet | 2

9. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure, respiratory rate, radial pulse and body temperature.
Time Frame: Screening up to Day 180 after last injection
Population: Safety set included all participants who received at least 1 injection of Xiapex.
Measure: Number; unit: participants
Arm/Group | Xiapex
Number analyzed (Participants) | 254
participants | 0

10. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid albumin, total protein); urinalysis (decimal logarithm of reciprocal of hydrogen ion activity [pH], glucose, protein, blood, ketones, microscopy[if urine tested positive for blood or protein]).
Time Frame: Screening up to Day 180 after last injection
Population: Safety set included all participants who received at least 1 injection of Xiapex.
Measure: Number; unit: participants
Arm/Group | Xiapex
Number analyzed (Participants) | 254
participants | 48

11. Other Pre Specified Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-clostridial type I collagenase (AUX-I) and anti-clostridial type II collagenase (AUX-II) antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Screening, Follow-up Day 180 after last injection
Population: Safety set included all participants who received at least 1 injection of Xiapex. 'Number of participants' analyzed signifies those participants who were evaluable for this outcome measure. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: participants
Arm/Group | Xiapex
Number analyzed (Participants) | 248
participants
  Screening: AUX-I Antibodies (n=248) | 6
  Screening: AUX-II Antibodies (n=248) | 3
  Follow-up Day 180: AUX-I Antibodies (n=239) | 220
  Follow-up Day 180: AUX-II Antibodies (n=239) | 215

12. Secondary Outcome: Number of Days of Concomitant Pain Medication Usage
Description: Amount of concomitant pain medication was assessed as the number of days participants used pain medication during the study.
Time Frame: Screening up to Day 180 after last injection
Population: Safety set included all participants who received at least 1 injection of Xiapex. 'Number of participants' analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Xiapex
Number analyzed (Participants) | 136
days | 2.0 [1 to 340]

13. Secondary Outcome: Number of Days Assessed on Dupuytren's Treatment Assessment Daily Diary Questionnaire
Description: Dupuytren's daily diary questionnaire assessed number of days during a cycle when 1) participant was absent or sick due to treatment, 2) the work hours were reduced, 3) the job duties were modified, 4) participant was unable to participate in hobbies and 5) participant wore a splint (for participants who were fitted for a splint).
Time Frame: C1D1 to C1D30, C2D1 to C2D30, C3D1 to C3D30, C4D1 to C4D30, C5D1 to C5D30
Population: FAS population. 'Number of participants' analyzed signifies those participants who were evaluable for this outcome measure. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Median (Full Range); unit: days
Arm/Group | Xiapex
Number analyzed (Participants) | 230
days
  C1D1 to C1D30: Absent or on sick leave (n=230) | 3.0 (3.80) [1 to 16]
  C1D1 to C1D30: Reduced work hours (n=230) | 2.0 (3.43) [1 to 16]
  C1D1 to C1D30: Modified job duties (n=230) | 2.0 (3.62) [1 to 16]
  C1D1 to C1D30: Not participated in hobbies (n=230) | 5.0 (4.61) [1 to 16]
  C1D1 to C1D30: Fitted with splint (n=211) | 12.0 (3.91) [1 to 16]
  C2D1 to C2D30: Absent or on sick leave (n=103) | 3.0 (3.33) [1 to 13]
  C2D1 to C2D30: Reduced work hours (n=103) | 2.0 (3.11) [1 to 12]
  C2D1 to C2D30: Modified job duties (n=103) | 2.0 (3.41) [1 to 12]
  C2D1 to C2D30: Not participated in hobbies (n=103) | 5.0 (4.61) [1 to 15]
  C2D1 to C2D30: Fitted with splint (n=96) | 11.0 (4.28) [1 to 16]
  C3D1 to C3D30: Absent or on sick leave (n=51) | 2.0 (4.53) [1 to 15]
  C3D1 to C3D30: Reduced work hours (n=51) | 3.0 (4.53) [1 to 14]
  C3D1 to C3D30: Modified job duties (n=51) | 3.0 (4.83) [1 to 14]
  C3D1 to C3D30: Not participated in hobbies (n=51) | 3.0 (5.05) [1 to 15]
  C3D1 to C3D30: Fitted with splint (n=44) | 10.0 (4.20) [1 to 15]
  C4D1 to C4D30: Absent or on sick leave (n=19) | 2.5 (3.61) [2 to 11]
  C4D1 to C4D30: Reduced work hours (n=19) | 2.0 (2.51) [1 to 7]
  C4D1 to C4D30: Modified job duties (n=19) | 2.0 (2.25) [1 to 7]
  C4D1 to C4D30: Not participated in hobbies (n=19) | 2.0 (3.75) [1 to 11]
  C4D1 to C4D30: Fitted with splint (n=15) | 10.5 (4.11) [4 to 16]
  C5D1 to C5D30: Absent or on sick leave (n=6) | 8.5 (4.95) [5 to 12]
  C5D1 to C5D30: Reduced work hours (n=6) | 8.5 (10.61) [1 to 16]
  C5D1 to C5D30: Modified job duties (n=6) | 10.5 (7.78) [5 to 16]
  C5D1 to C5D30: Not participated in hobbies (n=6) | 13.0 (6.22) [2 to 16]
  C5D1 to C5D30: Fitted with splint (n=5) | 11.0 (5.94) [1 to 16]

14. Secondary Outcome: Time to Recovery
Description: Time to recovery of normal activities was defined as median number of days between the initial injection date and the date on which participant recovered to normal activities, assessed after first, second and third injection for joints that received 1 through 3 injections. If a participant did not achieve recovery to normal activities, the participant's time to recovery was defined as the median number of days between the initial injection date and the date of the participant's the last daily diary recording within the cycle.
Time Frame: Up to Day 30 after first, second and third injection
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Xiapex
Number analyzed (Participants) | 230
days
  First injection (n=230) | 3.0 [3.0 to 4.0]
  Second injection (n=103) | 4.0 [2.0 to 5.0]
  Third injection (n=51) | 3.0 [2.0 to 4.0]

15. Secondary Outcome: Hand Functionality: Unite Rhumatologique Des Affections de la Main (URAM) Scale Total Score
Description: URAM:9-item questionnaire used to assess daily hand functionality.Participants rated their ability to perform following hand functionalities on 0 to 5 scale(0=without difficulty,5=impossible):1)washing themselves with flannel, keeping hand flat,2)washing face,3)holding bottle in one hand,4)shaking someone's hand,5)stroking/caressing someone,6)clapping,7)spreading out fingers, 8)leaning on hand,9)picking up small objects with thumb and index finger.URAM total score=sum of 9 items.Total score range=0 to 45,where higher score= higher difficulty in daily hand functionality.For each cycle, baseline value=pre-injection value reported at that cycle. For follow-up on Day 90,180 after last injection, baseline value (follow-up baseline)=pre-injection value reported at cycle 1. If response was provided to less than or equal to 4 items,URAM total score was considered missing. If response was provided to >=5 items, then average score of answered questions was imputed response to missing questions.
Time Frame: Baseline for cycle 1, 2, 3, 4, 5; C1D30, C2D30, C3D30, C4D30, C5D30; Follow-up Day 90, 180 after last injection
Population: as for outcome 13
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Xiapex
Number analyzed (Participants) | 126
units on a scale
  Baseline for cycle 1 (n=85) | 13.0 [0 to 32]
  C1D30 (n=89) | 3.0 [0 to 29]
  Baseline for cycle 2 (n=47) | 7.0 [0 to 36]
  C2D30 (n=51) | 4.0 [0 to 36]
  Baseline for cycle 3 (n=31) | 8.0 [0 to 36]
  C3D30 (n=31) | 3.0 [0 to 32]
  Baseline for cycle 4 (n=15) | 6.0 [0 to 32]
  C4D30 (n=15) | 5.6 [0 to 32]
  Baseline for cycle 5 (n=9) | 9.0 [0 to 32]
  C5D30 (n=9) | 2.3 [0 to 28]
  Baseline for Follow-up Day 90 (n=82) | 13.0 [0 to 32]
  Follow-up Day 90 (n=108) | 1.0 [0 to 29]
  Baseline for Follow-up Day 180 (n=83) | 13.0 [0 to 32]
  Follow-up Day 180 (n=126) | 0.5 [0 to 38]

16. Secondary Outcome: Number of Participants With Response Assessed on Dupuytren's Healthcare Resource Utilization (HCRU) Questionnaire
Description: Dupuytren's HCRU is a questionnaire used to assess healthcare usage in participants. Participants answered whether or not since their last visit they 1) had seen any doctor, 2) used any services (including physical or hand therapy, occupational therapy, home health care therapy), 3) were treated in emergency room, 4) had outpatient/day-case surgery, 5) were hospitalized, 6) had diagnostic/therapeutic procedures or tests performed, 7) were admitted in nursing home, 8) required aids/devices to assist in their daily functioning.
Time Frame: Baseline for cycle 1, 2, 3, 4, 5; C1D7, C1D30, C2D7, C2D30, C3D7, C3D30, C4D7, C4D30, C5D7, C5D30; Follow-up Day 90, 180 after last injection
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Xiapex
Number analyzed (Participants) | 254
participants
  Baseline cycle 1: Seen any doctor (n=254) | 10
  Baseline cycle 1: Received any therapy (n=254) | 0
  Baseline cycle 1:Treated in emergency room(n=254) | 1
  Baseline cycle 1: Outpatient surgery (n=254) | 2
  Baseline cycle 1: Hospitalization (n=254) | 0
  Baseline cycle 1: Diagnostic test (n=254) | 2
  Baseline cycle 1: In nursing home (n=254) | 0
  Baseline cycle 1: Required aids/devices (n=254) | 1
  C1D7: Seen any doctor (n=252) | 21
  C1D7: Received any therapy (n=252) | 12
  C1D7: Treated in emergency room (n=252) | 4
  C1D7: Outpatient surgery (n=252) | 9
  C1D7: Hospitalization (n=252) | 1
  C1D7: Diagnostic test (n=252) | 2
  C1D7: In nursing home (n=252) | 0
  C1D7: Required aids/devices (n=252) | 1
  C1D30: Seen any doctor (n=251) | 14
  C1D30: Received any therapy (n=251) | 7
  C1D30: Treated in emergency room (n=251) | 2
  C1D30: Outpatient surgery (n=251) | 3
  C1D30: Hospitalization (n=251) | 2
  C1D30: Diagnostic test (n=251) | 4
  C1D30: In nursing home (n=251) | 0
  C1D30: Required aids/devices (n=251) | 1
  Baseline cycle 2: Seen any doctor (n=111) | 4
  Baseline cycle 2: Received any therapy (n=111) | 1
  Baseline cycle 2:Treated in emergency room(n=111) | 0
  Baseline cycle 2: Outpatient surgery (n=111) | 1
  Baseline cycle 2: Hospitalization (n=111) | 0
  Baseline cycle 2: Diagnostic test (n=111) | 2
  Baseline cycle 2: In nursing home (n=111) | 0
  Baseline cycle 2: Required aids/devices (n=111) | 0
  C2D7: Seen any doctor (n=112) | 4
  C2D7: Received any therapy (n=112) | 4
  C2D7: Treated in emergency room (n=112) | 0
  C2D7: Outpatient surgery (n=112) | 3
  C2D7: Hospitalization (n=112) | 0
  C2D7: Diagnostic test (n=112) | 0
  C2D7: In nursing home (n=112) | 0
  C2D7: Required aids/devices (n=112) | 1
  C2D30: Seen any doctor (n=111) | 5
  C2D30: Received any therapy (n=111) | 3
  C2D30: Treated in emergency room (n=111) | 0
  C2D30: Outpatient surgery (n=111) | 1
  C2D30: Hospitalization (n=111) | 1
  C2D30: Diagnostic test (n=111) | 2
  C2D30: In nursing home (n=111) | 0
  C2D30: Required aids/devices (n=111) | 1
  Baseline cycle 3: Seen any doctor (n=51) | 1
  Baseline cycle 3: Received any therapy (n=51) | 0
  Baseline cycle 3:Treated in emergency room(n=51) | 0
  Baseline cycle 3: Outpatient surgery (n=51) | 0
  Baseline cycle 3: Hospitalization (n=51) | 0
  Baseline cycle 3: Diagnostic test (n=51) | 2
  Baseline cycle 3: In nursing home (n=51) | 0
  Baseline cycle 3: Required aids/devices (n=51) | 0
  C3D7: Seen any doctor (n=54) | 1
  C3D7: Received any therapy (n=54) | 0
  C3D7: Treated in emergency room (n=54) | 0
  C3D7: Outpatient surgery (n=54) | 1
  C3D7: Hospitalization (n=54) | 0
  C3D7: Diagnostic test (n=54) | 0
  C3D7: In nursing home (n=54) | 0
  C3D7: Required aids/devices (n=54) | 0
  C3D30: Seen any doctor (n=54) | 2
  C3D30: Received any therapy (n=54) | 1
  C3D30: Treated in emergency room (n=54) | 0
  C3D30: Outpatient surgery (n=54) | 1
  C3D30: Hospitalization (n=54) | 0
  C3D30: Diagnostic test (n=54) | 0
  C3D30: In nursing home (n=54) | 0
  C3D30: Required aids/devices (n=54) | 1
  Baseline cycle 4: Seen any doctor (n=23) | 1
  Baseline cycle 4: Received any therapy (n=23) | 0
  Baseline cycle 4:Treated in emergency room(n=23) | 0
  Baseline cycle 4: Outpatient surgery (n=23) | 0
  Baseline cycle 4: Hospitalization (n=23) | 0
  Baseline cycle 4: Diagnostic test (n=23) | 0
  Baseline cycle 4: In nursing home (n=23) | 0
  Baseline cycle 4: Required aids/devices (n=23) | 1
  C4D7: Seen any doctor (n=24) | 0
  C4D7: Received any therapy (n=24) | 2
  C4D7: Treated in emergency room (n=24) | 0
  C4D7: Outpatient surgery (n=24) | 0
  C4D7: Hospitalization (n=24) | 0
  C4D7: Diagnostic test (n=24) | 0
  C4D7: In nursing home (n=24) | 0
  C4D7: Required aids/devices (n=24) | 0
  C4D30: Seen any doctor (n=24) | 1
  C4D30: Received any therapy (n=24) | 1
  C4D30: Treated in emergency room (n=24) | 0
  C4D30: Outpatient surgery (n=24) | 0
  C4D30: Hospitalization (n=24) | 0
  C4D30: Diagnostic test (n=24) | 0
  C4D30: In nursing home (n=24) | 0
  C4D30: Required aids/devices (n=24) | 0
  Baseline cycle 5: Seen any doctor (n=12) | 0
  Baseline cycle 5: Received any therapy (n=12) | 0
  Baseline cycle 5:Treated in emergency room(n=12) | 0
  Baseline cycle 5: Outpatient surgery (n=12) | 0
  Baseline cycle 5: Hospitalization (n=12) | 0
  Baseline cycle 5: Diagnostic test (n=12) | 0
  Baseline cycle 5: In nursing home (n=12) | 0
  Baseline cycle 5: Required aids/devices (n=12) | 0
  C5D7: Seen any doctor (n=12) | 0
  C5D7: Received any therapy (n=12) | 0
  C5D7: Treated in emergency room (n=12) | 0
  C5D7: Outpatient surgery (n=12) | 0
  C5D7: Hospitalization (n=12) | 0
  C5D7: Diagnostic test (n=12) | 0
  C5D7: In nursing home (n=12) | 0
  C5D7: Required aids/devices (n=12) | 0
  C5D30: Seen any doctor (n=12) | 0
  C5D30: Received any therapy (n=12) | 0
  C5D30: Treated in emergency room (n=12) | 0
  C5D30: Outpatient surgery (n=12) | 0
  C5D30: Hospitalization (n=12) | 0
  C5D30: Diagnostic test (n=12) | 0
  C5D30: In nursing home (n=12) | 0
  C5D30: Required aids/devices (n=12) | 0
  Follow-up Day 90: Seen any doctor (n=247) | 10
  Follow-up Day 90: Received any therapy (n=247) | 8
  Follow-up Day 90:Treated in emergency room(n=247) | 8
  Follow-up Day 90: Outpatient surgery (n=247) | 11
  Follow-up Day 90: Hospitalization (n=247) | 4
  Follow-up Day 90: Diagnostic test (n=247) | 4
  Follow-up Day 90: In nursing home (n=247) | 1
  Follow-up Day 90:Required aids/devices(n=247) | 1
  Follow-up Day 180: Seen any doctor (n=249) | 4
  Follow-up Day 180: Received any therapy (n=249) | 3
  Follow-up Day 180:Treated in emergency room(n=249) | 8
  Follow-up Day 180: Outpatient surgery (n=249) | 9
  Follow-up Day 180: Hospitalization (n=248) | 6
  Follow-up Day 180: Diagnostic test (n=247) | 1
  Follow-up Day 180: In nursing home (n=248) | 0
  Follow-up Day 180: Required aids/devices (n=248) | 3

17. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using Dupuytren's Healthcare Resource Utilization (HCRU) Questionnaire
Description: Dupuytren's HCRU is a questionnaire used to assess healthcare usage in participants. Participants answered how many times since their last visit they 1) had seen any doctor, 2) used any services (including physical or hand therapy, occupational therapy, home health care therapy), 3) were treated in emergency room, 4) had outpatient/day-case surgery, 5) were hospitalized, 6) had diagnostic/therapeutic procedures or tests performed.
Time Frame: as for outcome 16
Population: FAS population. 'Number of participants' analyzed signifies those participants who were evaluable for this outcome measure. 'n' signifies those participants who were evaluable for this measure at given time points. Data for number of events was not analyzed for participants who responded that they did not perform the event.
Measure: Median (Full Range); unit: events
Arm/Group | Xiapex
Number analyzed (Participants) | 21
events
  Baseline cycle 1: Seen any doctor (n=10) | 1.0 [1 to 2]
  Baseline cycle 1: Treated in emergency room (n=1) | 2.0 [2 to 2]
  Baseline cycle 1: Outpatient surgery (n=2) | 1.0 [1 to 1]
  Baseline cycle 1: Diagnostic test (n=2) | 1.0 [1 to 1]
  C1D7: Seen any doctor (n=21) | 1.0 [1 to 3]
  C1D7: Received any therapy (n=12) | 1.0 [1 to 6]
  C1D7: Treated in emergency room (n=4) | 1.0 [1 to 1]
  C1D7: Outpatient surgery (n=8) | 1.0 [1 to 2]
  C1D7: Hospitalization (n=1) | 1.0 [1 to 1]
  C1D7: Diagnostic test (n=2) | 1.0 [1 to 1]
  C1D30: Seen any doctor (n=14) | 2.0 [1 to 4]
  C1D30: Received any therapy (n=7) | 2.0 [1 to 3]
  C1D30: Treated in emergency room (n=2) | 1.0 [1 to 1]
  C1D30: Outpatient surgery (n=3) | 1.0 [1 to 1]
  C1D30: Hospitalization (n=2) | 1.0 [1 to 1]
  C1D30: Diagnostic test (n=4) | 1.0 [1 to 2]
  Baseline cycle 2: Seen any doctor (n=4) | 1.0 [1 to 2]
  Baseline cycle 2: Received any therapy (n=1) | 1.0 [1 to 1]
  Baseline cycle 2: Outpatient surgery (n=1) | 1.0 [1 to 1]
  Baseline cycle 2: Diagnostic test (n=2) | 1.0 [1 to 1]
  C2D7: Seen any doctor (n=4) | 1.0 [1 to 2]
  C2D7: Received any therapy (n=3) | 1.0 [1 to 2]
  C2D7: Outpatient surgery (n=3) | 1.0 [1 to 1]
  C2D30: Seen any doctor (n=5) | 1.0 [1 to 13]
  C2D30: Received any therapy (n=3) | 4.0 [3 to 10]
  C2D30: Outpatient surgery (n=1) | 1.0 [1 to 1]
  C2D30: Hospitalization (n=1) | 1.0 [1 to 1]
  C2D30: Diagnostic test (n=2) | 1.0 [1 to 1]
  Baseline cycle 3: Seen any doctor (n=1) | 1.0 [1 to 1]
  Baseline cycle 3: Diagnostic test (n=2) | 1.0 [1 to 1]
  C3D7: Seen any doctor (n=1) | 1.0 [1 to 1]
  C3D7: Outpatient surgery (n=1) | 1.0 [1 to 1]
  C3D30: Seen any doctor (n=2) | 2.5 [2 to 3]
  C3D30: Received any therapy (n=1) | 1.0 [1 to 1]
  C3D30: Outpatient surgery (n=1) | 3.0 [3 to 3]
  Baseline cycle 4: Seen any doctor (n=1) | 2.0 [2 to 2]
  C4D7: Received any therapy (n=2) | 3.0 [3 to 3]
  C4D30: Seen any doctor (n=1) | 1.0 [1 to 1]
  C4D30: Received any therapy (n=1) | 6.0 [6 to 6]
  Follow-up Day 90: Seen any doctor (n=10) | 1.5 [1 to 3]
  Follow-up Day 90: Received any therapy (n=8) | 2.0 [1 to 45]
  Follow-up Day 90: Treated in emergency room (n=8) | 1.0 [1 to 2]
  Follow-up Day 90: Outpatient surgery (n=11) | 1.0 [1 to 3]
  Follow-up Day 90: Hospitalization (n=4) | 1.0 [1 to 1]
  Follow-up Day 90: Diagnostic test (n=4) | 1.0 [1 to 4]
  Follow-up Day 180: Seen any doctor (n=4) | 1.5 [1 to 3]
  Follow-up Day 180: Received any therapy (n=3) | 3.0 [2 to 22]
  Follow-up Day 180: Treated in emergency room (n=8) | 1.0 [1 to 3]
  Follow-up Day 180: Outpatient surgery (n=9) | 1.0 [1 to 5]
  Follow-up Day 180: Hospitalization (n=6) | 1.0 [1 to 2]
  Follow-up Day 180: Diagnostic test (n=1) | 1.0 [1 to 1]

18. Secondary Outcome: Number of Days as Assessed Using Dupuytren's Healthcare Resource Utilization (HCRU) Questionnaire
Description: Dupuytren's HCRU is a questionnaire used to assess healthcare usage in participants. Participants answered how many days since their last visit they 1) were hospitalized, 2) were in nursing home, 3) required aids/devices to assist in their daily functioning.
Time Frame: as for outcome 16
Population: FAS population. 'Number of participants' analyzed signifies those participants who were evaluable for this outcome measure. 'n' signifies those participants who were evaluable for this measure at given time points. Data for number of days was not analyzed for participants who responded that they did not perform the event.
Measure: Median (Full Range); unit: days
Arm/Group | Xiapex
Number analyzed (Participants) | 6
days
  Baseline cycle 1: Required aids/devices (n=1) | 8.0 [8 to 8]
  C1D7: Hospitalization (n=1) | 2.0 [2 to 2]
  C1D7: Required aids/devices (n=1) | 2.0 [2 to 2]
  C1D30: Hospitalization (n=2) | 8.5 [7 to 10]
  C1D30: Required aids/devices (n=1) | 20.0 [20 to 20]
  C2D7: Required aids/devices (n=1) | 8.0 [8 to 8]
  C2D30: Hospitalization (n=1) | 3.0 [3 to 3]
  C2D30: Required aids/devices(n=1) | 6.0 [6 to 6]
  C3D30: Required aids/devices (n=1) | 5.0 [5 to 5]
  Baseline cycle 4: Required aids/devices (n=1) | 5.0 [5 to 5]
  Follow-up: Day 90: Hospitalization (n=4) | 9.5 [2 to 21]
  Follow-up: Day 90: In nursing home (n=1) | 21.0 [21 to 21]
  Follow-up: Day 90: Required aids/devices(n=1) | 16.0 [16 to 16]
  Follow-up: Day 180: Hospitalization (n=6) | 2.5 [1 to 47]
  Follow-up: Day 180: Required aids/devices (n=1) | 2.0 [2 to 2]

19. Primary Outcome: Total Passive Extension Deficit (TPED) at Baseline for Second Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. Baseline value for second injection was the TPED value taken closest and prior to the administration of second injection. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Baseline for second injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 65
degrees | 45.0 [15 to 145]

20. Primary Outcome: Total Passive Extension Deficit (TPED) at Baseline for Third Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. Baseline value for third injection was the TPED value taken closest and prior to the administration of third injection. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Baseline for third injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 21
degrees | 40.0 [0 to 80]

21. Primary Outcome: Total Passive Extension Deficit (TPED) at Baseline for Fourth Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. Baseline value for fourth injection was the TPED value taken closest and prior to the administration of fourth injection. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Baseline for fourth injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 1
degrees | 20.0 [20 to 20]

22. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 1 After First Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 1 after first injection for fingers that received 1 injection. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 1 after first injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 256
degrees | 20.0 [0 to 165]

23. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 7 After First Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 7 after first injection for fingers that received 1 injection. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 7 after first injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 256
degrees | 10.0 [0 to 110]

24. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 30 After First Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 30 after first injection for fingers that received 1 injection. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 30 after first injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 257
degrees | 10.0 [0 to 110]

25. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 1 After Second Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 1 after second injection for fingers that received 2 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 1 after second injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 64
degrees | 29.0 [0 to 145]

26. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 7 After Second Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 7 after second injection for fingers that received 2 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 7 after second injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 65
degrees | 20.0 [0 to 155]

27. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 30 After Second Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 30 after second injection for fingers that received 2 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 30 after second injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 64
degrees | 20.0 [0 to 145]

28. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 1 After Third Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 1 after third injection for fingers that received 3 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 1 after third injection
Population: FAS: participants who received >= 1 injection of Xiapex, had >=1 post-injection efficacy assessment, whether goniometric or participant-reported. 'N' (number of participants analyzed) includes total number of participants in FAS, however actual 'N' for this outcome is unknown as these data were not calculated as per planned analysis.
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 19
degrees | 15.0 [0 to 70]

29. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 7 After Third Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 7 after third injection for fingers that received 3 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 7 after third injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 21
degrees | 22.0 [0 to 80]

30. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 30 After Third Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 30 after third injection for fingers that received 3 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 30 after third injection
Population: as for outcome 28
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 21
degrees | 30.0 [0 to 80]

31. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 1 After Fourth Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 1 after fourth injection for fingers that received 4 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 1 after fourth injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 1
degrees | 0.0 [0 to 0]

32. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 7 After Fourth Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 7 after fourth injection for fingers that received 4 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 7 after fourth injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 1
degrees | 0.0 [0 to 0]

33. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 30 After Fourth Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 30 after fourth injection for fingers that received 4 injections. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 30 after fourth injection
Population: as for outcome 28
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 1
degrees | 10.0 [10 to 10]

34. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 90 After Last Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 90 after the last injection, where last injection was a maximum up to fourth injection for a finger. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 90 after last injection
Population: as for outcome 2
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 244
degrees | 10.0 [0 to 120]

35. Primary Outcome: Total Passive Extension Deficit (TPED) at Day 180 After Last Injection
Description: TPED was defined as the sum of PED in the MP, PIP and DIP joints. PED was measured using finger goniometry. Passive extension=angle of the joint (MP or PIP or DIP) when the finger was passively extended as far possible toward the normal extension. PED=angle of deficit from normal extension. TPED was reported at Day 180 after the last injection, where last injection was a maximum up to fourth injection for a finger. 'Number of fingers/joints analyzed' signifies total number of fingers/joints that were evaluable for this outcome measure.
Time Frame: Day 180 after last injection
Population: as for outcome 28
Measure: Median (Full Range); unit: degrees
Units Other Than Participants: Fingers/Joints
Arm/Group | Xiapex
Number analyzed (Participants) | 254
Number analyzed (Fingers/Joints) | 250
degrees | 14.5 [0 to 195]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Xiapex
Serious Adverse Events (participants affected / at risk) | 12/254
Other Adverse Events (participants affected / at risk) | 212/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xiapex (N=254)
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Groin abscess (Infections and infestations) | 1
Groin infection (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Aortic valve disease mixed (Cardiac disorders) | 1
Transaminases increased (Investigations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dupuytren's contracture operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xiapex (N=254)
Lymphadenopathy (Blood and lymphatic system disorders) | 17
Lymph Node Pain (Blood and lymphatic system disorders) | 6
Oedema Peripheral (General disorders) | 111
Injection Site Pain (General disorders) | 53
Injection Site Haematoma (General disorders) | 39
Injection Site Swelling (General disorders) | 23
Injection Site Oedema (General disorders) | 20
Tenderness (General disorders) | 15
Axillary Pain (General disorders) | 10
Injection Site Vesicles (General disorders) | 10
Injection Site Haemorrhage (General disorders) | 9
Injection Site Erythema (General disorders) | 8
Malaise (General disorders) | 6
Nasopharyngitis (Infections and infestations) | 7
Skin Laceration (Injury, poisoning and procedural complications) | 37
Contusion (Injury, poisoning and procedural complications) | 34
Procedural Pain (Injury, poisoning and procedural complications) | 31
Surgical Skin Tear (Injury, poisoning and procedural complications) | 18
Post Procedural Swelling (Injury, poisoning and procedural complications) | 9
Post Procedural Complication (Injury, poisoning and procedural complications) | 8
Blood Glucose Increased (Investigations) | 6
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 65
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Joint Swelling (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6
Paraesthesia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 17
Pruritus (Skin and subcutaneous tissue disorders) | 13
Blood Blister (Skin and subcutaneous tissue disorders) | 12
Haematoma (Vascular disorders) | 49

LIMITATIONS AND CAVEATS:
Results were not reported for fifth injection as no finger received 5 injections.Results are reported for 'number of days of concomitant pain medication' as 'amount of pain medication' was interpreted as total number of days with pain medication use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.